CLINICAL TRIAL: NCT05291715
Title: The Effect of Ozone Therapy on Pain Perception After Free Gingival Graft Surgery in Patients With Mucogingival Defects A Randomized Controlled Clinical Trail
Brief Title: The Effect of Ozone Therapy on Pain Perception After Free Gingival Graft Surgery in Patients With Mucogingival Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omaima Mossad Mahmoud AL-Sherbini (Other)
Responsible Party: Sponsor-Investigator, Omaima Mossad Mahmoud AL-Sherbini, Principle investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 131221
Record Dates: First submitted 2022-02-22; First posted 2022-03-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Open Wound of Palate Without Complication; Pain, Postoperative; Free Gingival Grafts; Mucogingival Defects; Gingival Recession; Donor Site; Patient Satisfaction
Keywords: Ozone; Therapy; Pain; Gingival; Palatal; Donor; site; Recession; Mucogingival; Defects; Free; Grafts
MeSH Terms: conditions — Pain, Postoperative; Gingival Recession; Patient Satisfaction; Pain

STUDY DESIGN:
Intervention Model Description: Group 1: Will receive ozone therapy after harvesting a free gingival graft. Group 2: Following the harvesting of the free gingival graft; the palatal donor site will be protected by a periodontal pack.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double- blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1, test group (Experimental): This group will receive ozone therapy after harvesting of the free gingival graft from the palatal donor site.
  Interventions: Device: Ozone generator device (Ozone DTA-APOZAa-enterprize CO9-Taiwan, R.0.C)
- group 2, control group (No Intervention): Following harvesting of the free gingival graft, the palatal donor site ozone application will be simulated without starting of the ozone generator and the covered ( protected) by a periodontal pack.

INTERVENTIONS:
Device: Ozone generator device (Ozone DTA-APOZAa-enterprize CO9-Taiwan, R.0.C) — Gaseous ozone ( O3-triatomic oxygen) activates the neuroprotective systems, improve the blood circulation, oxygen delivery, stimulate the immunocompetent cells and enhance the release of growth factors. Moreover, ozone therapy showed to increase the quality of life post-operatively to a free gingival graft harvesting and decrease post-operative pain sensation ( Tasdemir et al, 2016)
  Arms: group 1, test group

SUMMARY:
Gaseous ozone (O3-triatomic oxygen) is the third-strongest oxidizing agent worldwide. It influences the cellular and the humoral immune system, by stimulating the proliferation of immunocompetent cells and the synthesis of immunoglobulin. Additionally; biologically active substances, such as interleukins, leukotrienes and prostaglandins which are beneficial in reducing inflammation and wound healing are orchestrated following ozone application. Given that after harvesting of a free gingival graft from the palatal donor site, healing occurs by secondary intention process; for patients with mucogingival conditions. The investigators will compare the natural process of healing at the donor site versus the healing process consecutive to ozone application; with the primary outcome is to evaluate the postoperative pain perception using visual analogue scale and to estimate the consumption of analgesics tablets after surgery.

DETAILED DESCRIPTION:
The procedures will be explained to all participants and they will be asked to sign an informed consent.

All patients will receive oral hygiene instructions and will receive phase I therapy comprising supragingival scaling and subgingival debridement.

After completion of phase I therapy the patients will be re-examined to ensure meeting all inclusion criteria. Then the participants will be allocated to 2 groups.

Group I will receive ozone therapy after harvesting free gingival graft. Group II following the harvesting of the free gingival graft, will be protected by a periodontal pack.

Surgical intervention:

Graft harvesting at donor site (Sullivan, & Atkins, 1968) To prepare the donor area, a rectangular-shape incision with 1-1.5 mm thickness will be made, and care will be taken to place most of the coronal part of the incision at least 2 mm apical from gingival margins of the upper teeth. The apical coronal dimension of the graft.

Following administration of anaesthesia by local infiltration (2% lidocaine with 1:100,000 epinephrine), a template will be placed over the palatal mucosa and will be used to outline the dimensions of the graft. The area chosen to harvest the free gingival graft will be chosen between first premolar and first molar.

The outlined graft will be carefully harvested as follows: The surgical blade entered in the contour incision, always in the posterior limit, sliding below the mucosa, and continued to find the opposite contour incision, in the anterior limit. The connective tissue surface will be carefully inspected for irregularities or adipose tissue after graft separation. Graft thickness will be immediately prepared (thinned) to obtain a graft approximately 1 to 1.5 mm thick.

The palatal wound will be protected by a periodontal pack; for the control group.

While the test group, will receive ozone therapy.

Ozone Application Protocol:

An ozone generator device (Ozone DTA-APOZAa- enterPrize Co9-Taiwan,R.0,C) with different probe numbers (#1 pointed probe,#2 pointed probe and #3 flat probe) will be used according to the manufacturer's instructions. Ozone will be applied on donor sites immediately after surgery and at days 1, 3, 7, 14 post-surgeries in the test group with output power at level 6-12 for 1 minute.

Ozone application in the control group will be simulated without starting the ozone generator.

Postoperative Protocol:

The participants will be instructed to abstain from brushing and flossing the teeth at the surgical area until suture removal (7days) and to use an antimicrobial rinse (0.12% chlorhexidine, 15 ml for 60 seconds twice daily) solution two times a day for 4 weeks.

The participants will be also instructed to consume only soft foods during the first week and to avoid any other mechanical trauma to the treated sites.

The participants will be given a prescription of Ibuprofen (600 mg every 12 hours) to be taken if necessary and the participants will be asked to record the number of tablets taken.

Participants will be enrolled in a professional plaque control program weekly for the first 4 weeks, then monthly until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects to be treated with free gingival grafts.
* Age older than 18 years old.
* No history of periodontal surgery in the area to be treated.
* Full mouth plaque score (FMPS) and full mouth bleeding score (FMBS) less than 20%.

Exclusion Criteria:

* Smoking
* Pregnancy and lactation.
* History of systematic diseases or medications that interferes with periodontal wound healing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of postoperative pain using visual analog scale. | 7 days
  Postoperative pain will be evaluated by visual analog scale (VAS) (Crichton, 2001).
  In this method, the patients will be asked to rate their pain at examination in form of a score between 0 (no pain) and 10 (the most pain which patient has ever experienced).
  This assessment will be made every day for the first 7 days following the FGG operation.
Evaluation of postoperative pain | 7 days
  The participants will report the number of analgesic tablets ingested to relieve the pain.

SECONDARY OUTCOMES:
Evaluation of complete epithelialization of the palatal wound. | 28 days
  Hydrogen peroxide test (H 2 O 2) for assessment of epithelialization in control and test groups and at days 7, 14, 21 and 28, a 3% H 2 O 2 will be sprinkled on the palatal wounds by using a syringe. If the epithelium is discontinuous, it diffuses into the connective tissue, and the enzyme catalase acts on H 2 O 2 to release water and oxygen showing bubbles on the wound of FGG. Complete epithelialization will be scored clinically, following visual inspection (Yes, no). If the epithelial barrier is intact, then H2O2 does not diffuse into the connective tissue, it is not acted upon by catalase, and oxygen is not liberated. Absence of bubble formation following hydrogen peroxide application will be scored as positive complete epithelialization (Silva et al.,2010).

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Professor of Oral Diagnosis,Oral Medicine and Periodontology Faculty of Dentistry,Cairo University.
Locations (1):
- Cairo University-Faculty of Dentistry, Cairo, Manial, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
The shared measures; clinical parameters will be shared pain perception by VAS scale, complete epitheliazation, evaluation of soft tissue healing at donor site.

REFERENCES:
- [Background] Miller PD Jr. Root coverage using the free soft tissue autograft following citric acid application. III. A successful and predictable procedure in areas of deep-wide recession. Int J Periodontics Restorative Dent. 1985;5(2):14-37. No abstract available. PMID 3858263
- [Background] Ozcan M, Ucak O, Alkaya B, Keceli S, Seydaoglu G, Haytac MC. Effects of Platelet-Rich Fibrin on Palatal Wound Healing After Free Gingival Graft Harvesting: A Comparative Randomized Controlled Clinical Trial. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):e270-e278. doi: 10.11607/prd.3226. PMID 28817141